CLINICAL TRIAL: NCT02202226
Title: Interventional, Randomised, Double-blind, Placebo-controlled, Sequential Group, Multiple Dose Study Investigating the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of Lu AF35700 in Patients With Schizophrenia
Brief Title: Safety and Tolerability Study of Lu AF35700 After Repeated Dosing in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14754A
Record Dates: First submitted 2014-07-25; First posted 2014-07-28 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lu AF35700

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lu AF35700 oral solution (1 mg/mL) (Experimental): Planned daily doses range from 5 mg/day to 30 mg/day for 3 weeks. Weekly doses up to 75 mg/week for 3 weeks.
  Interventions: Drug: Lu AF35700
- Matching placebo (Placebo Comparator): Oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AF35700
  Arms: Lu AF35700 oral solution (1 mg/mL)
Drug: Placebo
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of Lu AF35700 after repeated oral dosing to patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 60 years (extremes included)
* BMI of ≤38
* Primary diagnosis of schizophrenia according to DSM-IV-TR™ (codes 295.10, 295.20, 295.30, 295.90)
* Clinical Global Impression - Severity of Illness (CGI-S) score ≤4 (moderately ill) at screening and baseline
* PANSS total score ≤80
* Score ≤4 (moderate) on the following PANSS items at screening and safety baseline: P7 (hostility), G8 (uncooperativeness)
* Willing to be hospitalised for 4 to 5 weeks after the Safety Baseline Visit

Exclusion Criteria:

* The patient experienced an acute exacerbation requiring hospitalization within the last 6 months
* The patient experienced an acute exacerbation requiring change in antipsychotic medication (with reference to drug or dose) within the last 4 weeks
* The patient has a diagnosis or history of substance dependence (except nicotine) or substance abuse according to DSM-IV-TR® criteria ≤3 months prior to screening
* The patient smokes >20 cigarettes per day

Other protocol-defined inclusion and exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Absolute values and change from baseline in safety variables (Adverse events, clinical safety laboratory tets, vital signs, weight, and ECG) | Screening to day 78 (up to 8 weeks after last dose)
Change from baseline in AIMS, BARS and SAS Total score | Baseline to day 21
  Abnormal movement rating scale
Columbia Suicide Severity Rating Scale (C-SSRS) | Sceening to day 78 (up to 8 weeks after last dose)

SECONDARY OUTCOMES:
Day 21 area under the Lu AF35700 and Lu AF36152 plasma concentration-time curve from 0-24 hours post dose (AUC0-tau) in a daily dosing regime | Day 21 in the dosing period
Maximum observed concentration (Cmax) of Lu AF35700 and Lu AF36152 | Day 1 and 21 in the dosing period
Half-lives (t½) of Lu AF35700 and Lu AF36152 | Day 1 and 21 in the dosing period
Day 14-21 area under the Lu AF35700 and LuAF36152 plasma-concentration-time curve from 0-168 hours post-dose (AUCtau) in a weekly dosing regimen | Day 14-21 in the dosing period

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H.Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- PAREXEL Phase I Unit, Glendale, California, United States